CLINICAL TRIAL: NCT04520230
Title: Comparative Study Between Three Therapeutic Options for Treatment of Chronic Obstructive Pulmonary Disease Patients
Brief Title: Three Treatment of Chronic Obstructive Pulmonary Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dr. Tarek Mohamed Mostafa, Associate Professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP00011
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination; Tiotropium Bromide; Formoterol Fumarate

STUDY DESIGN:
Intervention Model Description: randomized double blind prospective study.
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Group 1: 15 patients with COPD who will receive inhaled corticosteroid (ICS)plus long acting B2-agonist (LABA) (Budesonide/Formoterol combination (160/4.5mcg) 2 inhalations bid).
  Interventions: Drug: Budesonide/Formoterol combination 160/4.5 mcg, 2 inhalations bid
- Group 2 (Experimental): Group 2: 15 patients with COPD who will receive inhaled corticosteroid (ICS) plus long acting anticholinergic (LAAC) (Tiotropium 18 mcg inhaled capsule once daily+ Budesonide inhalation 200 mcg twice daily).
  Interventions: Drug: Tiotropium 18 mcg capsule inhaled once daily + Budesonide
- Group 3 (Experimental): Group 3: 15 patients with COPD who will receive long acting B2-agonist (LABA) plus long acting anticholinergic (LAAC). (Tiotropium 18 mcg inhaled capsule once daily+ Formoterol 12 mcg inhaled capsule twice daily)
  Interventions: Drug: Formoterol/Tiotropium

INTERVENTIONS:
Drug: Budesonide/Formoterol combination 160/4.5 mcg, 2 inhalations bid — inhaled corticosteroid (ICS)plus long acting B2-agonist (LABA) (Budesonide/Formoterol combination 160/4.5 mcg, 2 inhalations bid ).
  Other Names: Budesonide/Formoterol
  Arms: Group 1
Drug: Tiotropium 18 mcg capsule inhaled once daily + Budesonide — inhaled corticosteroid (ICS) plus long acting anticholinergic (LAAC) (Tiotropium 18 mcg capsule inhaled once daily + Budesonide ).
  Other Names: Tiotropium/ Budesonide
  Arms: Group 2
Drug: Formoterol/Tiotropium — long acting B2-agonist (LABA) plus long acting anticholinergic (LAAC).
  Other Names: LABA /LAAC.
  Arms: Group 3

SUMMARY:
Forty five COPD patients will be recruited from Chest Disease Department, Tanta University Hospital, Tanta, Egypt.

The aim of the study is to Compare between the effectiveness of three therapeutic options for treatment of moderate and severe COPD patients .These therapeutic options include Inhaled corticosteroid (ICS) plus long acting B2-agonist (LABA) combination, Inhaled corticosteroid (ICS) plus long acting anticholinergic (LAAC) combination and Long acting B2-agonist (LABA) plus long acting anticholinergic (LAAC) combination .

DETAILED DESCRIPTION:
This study will be prospective randomized double blind study.

The forty five COPD patients will be divided into three groups:

Group 1: 15 patients with COPD who will receive inhaled corticosteroid (ICS)plus long acting B2-agonist (LABA) (Budesonide/Formoterol combination 160/4.5 mcg, 2 inhalations bid ).

Group 2: 15 patients with COPD who will receive inhaled corticosteroid (ICS) plus long acting anticholinergic (LAAC) (Tiotropium 18 mcg capsule inhaled once daily + Budesonide ).

Group 3: 15 patients with COPD who will receive long acting B2-agonist (LABA) plus long acting anticholinergic (LAAC).

If any worsening of dyspnea, increase of purulence, or increase of sputum production appear plus increase of peak variability more than 35% and FEV1 that necessitate a change of the regular drug medication of the patient will be recorded as exacerbation.

All patients will be submitted to the following analysis at the baseline, during and 12 weeks after the assigned treatment:

1. Full medical history will be taken through clinical assessment of dyspnea, chronic cough and sputum production using mMRC or CAT test.
2. Forced expiratory volume in 1second (FEV1) value measurement using spirometry.
3. Measurement of the following inflammatory markers in serum and/ or plasma of patients under study .

   * Tumer necrosis factor alpha ( TNF )
   * Fibrinogen
   * Interlukin 6 ( IL6 )

Statistical analysis

The results will be statistically calculated to evaluate its clinical significance if any before ,during and after drug therapy using (ANOVA) system SPSS version 20 (2012) to compare between the three groups of patients and paired t-test will be used to compare between results before, during and after drug therapy .

ELIGIBILITY:
Inclusion Criteria:

1. Age from 30 to 40 years or older.
2. Patient with 30%≥ FEV1<80% predicted and FEV1/FVC <70% predicted.

Exclusion Criteria:

1. Patients with FEV1< 30% predicted or FEV1< 50% predicted plus chronic respiratory failure.
2. Patients with recent chest infection or had been hospitalised for an exacerbation or respiratory infection in the 6 weeks before screening.
3. Patients with history of asthma.
4. Patient with clinically significant condition ex; unstable ischemic heart disease, uncontrolled hypertension, uncontrolled diabetes.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
FEV1 value | three months
  Forced expiratory volume in 1second (FEV1) value
Tumer necrosis factor alpha ( TNF ) | three months
  serum level
Interlukin 6 ( IL6 ) | three months
  serum level
Fibrinogen | Three months
  serum level

CONTACTS AND LOCATIONS:
Overall Officials: Tarek M Mostafa, Ass. Prof., Principal Investigator — Tanta University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qaseem A, Wilt TJ, Weinberger SE, Hanania NA, Criner G, van der Molen T, Marciniuk DD, Denberg T, Schunemann H, Wedzicha W, MacDonald R, Shekelle P; American College of Physicians; American College of Chest Physicians; American Thoracic Society; European Respiratory Society. Diagnosis and management of stable chronic obstructive pulmonary disease: a clinical practice guideline update from the American College of Physicians, American College of Chest Physicians, American Thoracic Society, and European Respiratory Society. Ann Intern Med. 2011 Aug 2;155(3):179-91. doi: 10.7326/0003-4819-155-3-201108020-00008. PMID 21810710
- [Background] Falk JA, Minai OA, Mosenifar Z. Inhaled and systemic corticosteroids in chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2008 May 1;5(4):506-12. doi: 10.1513/pats.200707-096ET. PMID 18453363
- [Derived] Mostafa TM, El-Azab GA, Atia GA, Lotfy NS. The Effectiveness of 3 Combined Therapeutic Regimens in Egyptian Patients with Moderate-to-Severe Chronic Obstructive Pulmonary Disease: A Randomized Double-Blind Prospective Pilot Study. Curr Ther Res Clin Exp. 2021 Mar 8;94:100625. doi: 10.1016/j.curtheres.2021.100625. eCollection 2021. PMID 34306265